CLINICAL TRIAL: NCT02916017
Title: HUMIRA® Special Investigation (Long-term Treatment in Patients With Non-infectious Intermediate-, Posterior-, or Pan-uveitis)
Brief Title: HUMIRA® Long-term Treatment in Patients With Non-infectious Intermediate-, Posterior-, or Pan-uveitis
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P15-665
Record Dates: First submitted 2016-09-14; First posted 2016-09-27 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Uveitis
Keywords: Humira; Adalimumab; Non-infectious Intermediate-, Posterior-, or Pan-uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants receiving adalimumab: Participants receiving adalimumab for the treatment of Non-infectious Intermediate-, Posterior-, or Pan-uveitis

SUMMARY:
This study evaluates the long- term safety and effectiveness of adalimumab in participants with non-infectious intermediate-, posterior-, or pan-uveitis in daily practice in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Participants receiving adalimumab for the treatment of Non-infectious Intermediate-, Posterior-, or Pan-uveitis

Exclusion Criteria:

* Participants previously treated with adalimumab

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Non-infectious Intermediate-, Posterior-, or Pan-uveitis
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-10-14 (Actual); Study Completion 2020-10-14 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADR) | Up to Week 52
  ADR is the causal relationship between adalimumab and adverse events.

SECONDARY OUTCOMES:
Change in Visual Functioning Questionnaire (VFQ)-25 score | From Week 0 (baseline) to Week 52
  The National Eye Institute VFQ-25 is an ocular disease-specific survey that measures the influence of visual disability and visual symptoms on generic health domains such as emotional well-being and social functioning, in addition to task-oriented domains related to daily visual functioning. The VFQ-25 consists of a base set of 25 vision-targeted questions plus an additional single-item general health rating question. The overall composite score ranges from 0 to 100, where higher scores or increases in score indicate better vision-related functioning.
Change in Visual acuity in each eye | From Week 0 (baseline) to Week 52
  Visual acuity change is assessed.
Change in Anterior Chamber (AC) cell grade (standardization of uveitis nomenclature (SUN) criteria) in each eye | From Week 0 (baseline) to Week 52
  Slit lamp examinations will be conducted at each visit to assess AC cell count. The number of AC cells observed within a 1 mm × 1 mm slit beam will be used to determine the grade according to the Standardization of Uveitis Nomenclature (SUN) criteria:
  Grade 0 = < 1 cell
  Grade 0.5+ = 1 - 5 cells
  Grade 1+ = 6 - 15 cells
  Grade 2+ = 16 - 25 cells
  Grade 3+ = 26 - 50 cells
  Grade 4+ = > 50 cells.
Percentage of Overall improvement | Up to Week 52
  This is assessed by physicians.
Change in retinal lesions in each eye | From Week 0 (baseline) to Week 52
  The change in retinal lesion are assessed.
Change in central retinal thickness in each eye | From Week 0 (baseline) to Week 52
  This is assessed by Optical Coherence Tomography (OCT)
Change in Vitreous Haze grade in each eye | From Week 0 (baseline) to Week 52
  Vitreous haze will be measured using dilated indirect ophthalmoscopy (DIO) and assessed by the Investigator according to National Eye Institute (NEI)/ SUN criteria:
  Grade 0: No evident vitreous haze;
  Grade 0.5+: Slight blurring of the optic disc margin because of the haze; normal striations and reflex of the nerve fiber layer cannot be visualized;
  Grade 1+: Permits a better definition of both the optic nerve head and the retinal vessels (compared to higher grades);
  Grade 2+: Permits better visualization of the retinal vessels (compared to higher grades);
  Grade 3+: Permits the observer to see the optic nerve head, but the borders are quite blurry;
  Grade 4+: Optic nerve head is obscured.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (39):
- Japan (39):
  - Juntendo University Urayasu Hospital /ID# 168358, Urayasu-shi, Chiba
  - Matsuyama Red Cross Hospital /ID# 164149, Matsuyama, Ehime
  - Kyushu University Hospital /ID# 163042, Fukuoka, Fukuoka
  - Fukuoka University Hospital /ID# 163043, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 162945, Kurume-shi, Fukuoka
  - Gunma University Hospital /ID# 166916, Maebashi, Gunma
  - Hiroshima University Hospital /ID# 166915, Hiroshima, Hiroshima
  - Hokkaido University Hospital /ID# 163041, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 165250, Kobe, Hyōgo
  - Duplicate_Kanazawa University Hospital /ID# 166914, Kanazawa, Ishikawa-ken
  - Yokohama Municipal Citizen's Hospital /ID# 161742, Yokohama, Kanagawa
  - Kochi Medical School Hospital /ID# 164144, Nankoku-shi, Kochi
  - Shinshu University Hospital /ID# 164153, Matsumoto-shi, Nagano
  - Niigata University Medical & Dental Hospital /ID# 169563, Niigata, Niigata
  - Osaka University Hospital /ID# 164147, Suita-shi, Osaka
  - Saitama Medical University Hospital /ID# 162944, Iruma-gun, Saitama
  - Dokkyo Medical University Hospital /ID# 164154, Shimotsuga-gun, Tochigi
  - Tokushima University Hospital /ID# 164145, Tokushima, Tokushima
  - Juntendo University Hospital /ID# 169564, Bunkyo-ku, Tokyo
  - Tokyo Medical And Dental University, Medical Hospital /ID# 165251, Bunkyo-ku, Tokyo
  - Nippon Medical School Hospital /ID# 166938, Bunkyo-ku, Tokyo
  - The University of Tokyo Hospital /ID# 162943, Bunkyo-ku, Tokyo
  - The Jikei University Hospital /ID# 164152, Minato-ku, Tokyo
  - Tokyo Medical University Hospital /ID# 164146, Shinjuku-ku, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine /ID# 164148, Shinjuku-ku, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 165248, Shinjuku-ku, Tokyo
  - Yamaguchi University Hospital /ID# 165249, Ube-shi, Yamaguchi
  - Kagoshima Uni Med and Dental /ID# 164150, Kagoshima
  - Kakogawa Central City Hospital /ID# 167706, Kakogawa
  - Miyata Ophthalmic Hospital /ID# 167707, Miyakonojō
  - Duplicate_The Hospital of Hyogo College /ID# 166913, Nishinomiya-shi
  - Osaka Hospital /ID# 164151, Osaka
  - Yodogawa Christian Hospital /ID# 161741, Osaka
  - Omihachiman Community Med Ctr /ID# 164978, Ōmihachiman
  - Tosei General Hospital /ID# 167708, Seto
  - Natl Defense Med College Hosp /ID# 162946, Tokorozawa
  - Abbott Japan /ID# 147893, Tokyo
  - Tokyo Shinjuku Medical Center /ID# 166934, Tokyo
  - Tottori Municipal Hospital /ID# 159431, Tottori

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Namba K, Kaburaki T, Tsuruga H, Ogawa Y, Iwashita E, Goto H. Long-Term Safety and Effectiveness of Adalimumab in Japanese Patients with Noninfectious Intermediate, Posterior, or Panuveitis: Post-Marketing Surveillance of 251 Patients. Ophthalmol Ther. 2022 Jun;11(3):1147-1161. doi: 10.1007/s40123-022-00493-z. Epub 2022 Mar 19. PMID 35305254
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/adalimumab_P15-665.pdf